CLINICAL TRIAL: NCT05313581
Title: Implementation of an E-version of the Skills Training START NOW for Promoting Emotion Regulation and Resilience in Residential Youth Care and Correctional Institutions: a Cluster Randomized Controlled Trial
Brief Title: START NOW WebApp: Skill Training for Promoting Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Christina Stadler (Network)
Responsible Party: Sponsor-Investigator, Prof. Christina Stadler, Principal Investigator, Professor for Developmental Psychopathology (Full professorship), Department of Child and Adolescent Psychiatry (UPK-KJ), Psychiatric University Clinics Basel (UPK), University Psychiatric Clinics Basel
Organization: University Psychiatric Clinics Basel (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-00108
Record Dates: First submitted 2022-03-16; First posted 2022-04-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Resilience; Emotion Regulation; Social Competence; Stress
MeSH Terms: conditions — Emotional Regulation; Social Skills

STUDY DESIGN:
Intervention Model Description: 1) Web-based group training guided by a trained START NOW facilitator(either face-to-face or through videoconferencing)2) Web-based self-help without guidance 3) Treatment as usual (TAU)
Masking Description: open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- START NOW as web-based group training guided by a facilitator (Active Comparator): In condition 1, participants will be required to attend weekly sessions of the group training (period of 9 weeks; 3 double sessions;4 to12 participants) guided by a facilitator, either face-to-face or via videoconferencing. Facilitation will be provided either by a staff member (caretaker) of the institution who has received a 1.5 days training in START NOW (face-to-face setting), or by a member of the START NOW facilitator team of Universitäre Psychiatrische Kliniken (UPK) Basel (videoconference setting). All participants will have access to the START NOW Web application (WebApp) during the entire intervention and follow-up phase to complete additional exercises or review content.
  Institutions randomized to group training guided by a facilitator condition will receive the complete pretraining (12 hours à 3 blocks: Theoretical Background; WebApp and Facilitator Material; Running Sessions) with individual coaching. Supervision will be provided twice during the intervention phase.
  Interventions: Behavioral: START NOW WebApp
- START NOW as web-based pure self-help training (Active Comparator): Participants in condition 2 will use the START NOW web-based pure self-help training. Using the same session contents as in the group training guided by a facilitator, sessions have been adjusted so that participants can complete them individually and participants receive one session each week (session 1+2, 9+10 and 11+12 as double sessions). Institutions randomized to pure self-help training will receive the first block of the pretraining and the material from the second block (facilitator training material) prior to interventions start.
  Interventions: Behavioral: START NOW WebApp
- Treatment as usual (TAU) (No Intervention): Participants in condition 3 will not receive any health promotion services during the skills training or follow-up period beyond what is offered at their respective institution. They will also be excluded from any group trainings similar to START NOW. For ethical reasons and to increase study-related commitment, they will be provided with the web-based pure self-help training after completion of the study. Institution staff will receive the first block of the pretraining and material from the second block after the end of the intervention. Supervision for participating caretakers and facilitators will not be provided during the intervention phase.

INTERVENTIONS:
Behavioral: START NOW WebApp — The WebApp is based on the existing manualized START NOW skills training. START NOW aims to improve emotion- and stress regulation, social competence, effective management of encountered problems/crises, subjective well-being and resilience through improving an individual's level of psychological flexibility. It primarily employs a cognitive behaviourally oriented group skills training with integrated components from Dialectical Behavioural Therapy (DBT), Acceptance and Commitment Therapy (ACT), trauma-informed care and Motivational Interview (MI) techniques.
  During the training, participants will encounter different exercises to help them train their skills. There are several mindfulness exercises in the form of audio tracks, containing, e.g., instructions on a breathing exercise. The skills training phase takes place over a period of 9 weeks (sessions 1+2, 9+10 and 11+12 are double session).
  Arms: START NOW as web-based group training guided by a facilitator; START NOW as web-based pure self-help training

SUMMARY:
Almost every young person has experienced difficult situations, crises and stress in his or her life. It is difficult to cope with such situations and it is not uncommon for mental health to be affected. At the same time, those affected often do not get any help. There are too few offers of help. That is why the investigators have developed the START NOW training and the corresponding WebAPP. With this training, young people can train their resilience, i.e. their psychological resistance. Resilient people cope better with difficult situations and remain psychologically healthy for longer. Because the START NOW training is now also available as a WebAPP, users can apply it practically, playfully and at any time. Furthermore, the WebAPP can be used as a prevention and treatment option in a resource-saving and cost-efficient way in institutions. The aim is to find out in a randomized study design with two treatment conditions and a waiting group whether START NOW is effective as a newly developed WebAPP. Specifically, the investigators will investigate whether a digital web-based self-help training can already achieve positive effects or whether a format in which accompanying guidance by a coach and social learning is possible (support by a trainer who guides young people during the training) is better for achieving sustainable changes.The project is funded by the Federal Office of Justice as part of a pilot project.

DETAILED DESCRIPTION:
Psychological Flexibility (PF) is associated with improved mental health across a multitude of contexts and populations, while psychological inflexibility is associated with mental health problems, in particular depression and anxiety. Taking into consideration that prevalence rates of clinically significant anxiety and depression in large youth cohorts are high and even increased especially due to Covid-19, interventions aiming to enhance psychological flexibility are of particular importance. START NOW represents one approach that is well equipped to promote PF. It is an evidence-based, integrative skills training program, which offers a broad scope of applicability to different populations and contexts by promoting general psychological health and resilience.

Web-based health approaches are well established across settings, populations and a range of mental health outcomes and offer benefits such as cost-effectiveness, high accessibility and flexibility, direct and convenient use of resources, anonymity, decreased stigmatization and a feasible way to ensure continuity of care in transitional phases. Our project aims to develop and evaluate a web-based translation of the existing START NOW skills training that promotes PF in institutionalized youth.

The investigatorss will investigate the efficacy of web-based START NOW on PF in a randomized controlled trial comparing the following conditions: 1) Web-based group training guided by a trained START NOW facilitator (either face-to-face or through videoconferencing) 2) Web-based self-help without guidance 3) Treatment as usual (TAU)

ELIGIBILITY:
Inclusion Criteria:

* Youth and young adults in Residential Youth Care (RYC) or Correctional Institutions (CI)
* Age between 14-24 at time of screening
* Need for improvement: Avoidance and Fusion Questionnaire for Youth (AFQ-Y) equal or higher than 34.05, or
* Massachusetts Youth Screening Instrument-2 (MAYSI-2) subscale Angry-Irritable equal or higher than 5, or
* MAYSI-2 subscale Depressed-Anxious equal or higher than 3.
* Sufficient speaking, writing and reading skills in German or French
* (Written) informed consent
* No planned discharge before end of intervention phase; Exception: Self-Help condition

Exclusion Criteria:

* Suicidality: MAYSI-2 subscale Suicide Ideation equal or higher than 2
* Acute psychotic symptoms or mania: MAYSI-2 subscale Thought Disturbance equal or higher than 1
* Concurrent Cognitive Behavioral Therapy (CBT) based skills training similar to START NOW

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Response to web-based training: pre-post participation CHANGE in psychological inflexibility as measured by scores on the AFQ-Y questionnaire | Primary endpoint is the CHANGE in total score between baseline (T1) and follow-up (T3, 12 +/- 2 weeks after the end of the intervention)
  The AFQ-Y is a widely used and validated self-rating questionnaire for assessing Psychological Flexibility in youth and young adults. Participants answer 17 items indicating how true each item is for them on a 5-point Likert scale (0 = not at all true; 4 = very true). Higher total scores indicate lower PF. Items are based on ACT models of human suffering representing the theoretical concept of psychological inflexibility due to high cognitive fusion and experiential avoidance. Data will be assessed within 2 weeks before start of skills training (baseline, T1), within 2 weeks after end of skills training (post-treatment assessment, T2), as well as at 12 weeks (+/- 2 weeks) (T3) and 24 weeks (+/- 2 weeks) (T4) post skills training. Primary endpoint is the change in total score between baseline (T1) and follow-up (T3). Total scores can range between 0 and 68. Accordingly, a change in score can range between -68 to +68.

SECONDARY OUTCOMES:
change in resilience (all 3 conditions) | - between baseline (T1) and post-training (T2, ≤2 weeks after end of intervention ) - between baseline (T1) and 12-week follow-up (T3, after the end of intervention) - between baseline (T1) and 24-week follow-up (T4)
  Increase in total score on the German version of the Connor-Davidson Resilience Scale (CD-RISC) in the 10-items version both in self-rating by participant and self-rating by caretaker. The CD-RISC refers to an individual's ability to endure difficult experiences. Answers are given on a 5-point Likert-Scale (0= not true at all; 4= true nearly all of the time). Total scores can range from 0 to 50, with change scores ranging from -50 to +50.
change in self-reported psychological well-being (all 3 conditions) | - between baseline (T1) and post-training (T2, ≤2 weeks after end of intervention ) - between baseline (T1) and 12-week follow-up (T3, after the end of intervention) - between baseline (T1) and 24-week follow-up (T4)
  Increase in total score on the World Health Organization - Five Well-Being Index (WHO-5) in self-rating by participant. The self-report questionnaire contains five items on a 6-point Likert-Scale (5= all of the time; 0= none of the time). Respondents are asked to indicate how often they felt well during the last two weeks. Total scores can range from 0 to 25, with higher scores indicating greater well-being. Accordingly, change scores range from -25 to +25.
change in self-reported self-efficacy (all 3 conditions) | - between baseline (T1) and post-training (T2, ≤2 weeks after end of intervention ) - between baseline (T1) and 12-week follow-up (T3, after the end of intervention) - between baseline (T1) and 24-week follow-up (T4)
  Increase in total score on the German 'General Self-Efficacy Scale - Skala zur Allgemeinen Selbstwirksamkeitserwartung' (SWE) in self-rating by participant. The questionnaire includes 10 Items and a 4-point Likert Scale (1= not true; 4= completely true). The scale reflects one's convictions on subjective controllability or competence expectations in different demand situations, with higher scores indicating a greater sense of self-efficacy. Total scores can range from 10 to 40, with change scores ranging from -40 to +40.
change in general impairment (all 3 conditions) | - between baseline (T1) and post-training (T2, ≤2 weeks after end of intervention ) - between baseline (T1) and 12-week follow-up (T3, after the end of intervention) - between baseline (T1) and 24-week follow-up (T4)
  Reduction of all sub scores and total score on the Columbia Impairment Scale (CIS) both in self-rating by participant and external rating by caretaker. The 13-item questionnaire captures functional impairment in four domains: interpersonal relations, broad psychopathological domains, functioning in school or at work, and use of leisure time. It will be answered both by the participant as a self-report questionnaire, and by the caretakers as external raters. Items are answered on a 5-point Likert-Scale (0= no problem; 4= a very big problem). Total score can range from 0 to 52, with change scores ranging from -52 to +52.
change in depression and anxiety (all 3 conditions) | - between baseline (T1) and post-training (T2, ≤2 weeks after end of intervention ) - between baseline (T1) and 12-week follow-up (T3, after the end of intervention) - between baseline (T1) and 24-week follow-up (T4)
  Reduction of total score on the Patient Health Questionnaire 4 (PHQ-4) in self-rating by participants. The PHQ-4 is a ultra- short questionnaire with the two subscales depression and anxiety, and was evaluated a s a reliable, valid and precise screening tools for self reported depression, anxiety and general psychological distress. Answers are given on 4-point Likert-Scale (0=not at all, 3= nearly every day). Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.
change in anger-irritability (all 3 conditions) | - between baseline (T1) and post-training (T2, ≤2 weeks after end of intervention ) - between baseline (T1) and 12-week follow-up (T3, after the end of intervention) - between baseline (T1) and 24-week follow-up (T4)
  Reduction of total score on Affective Reactivity Scale (ARI) both in self-rating by participant and external rating by caretaker. The ARI contains seven items to be scored on a 3-point Likert-Scale (0= not true, 1= somewhat true, 2= certainly true). As just the first six items are summed to the total score, it can range from 0 to 12, with change scores ranging from -12 to +12. The seventh item is analysed separately.
change in substance use (all 3 conditions) | between screening (T0) and 12 week follow-up (T3, 12 weeks after the end of the intervention)
  Reduction of total score on the Alcohol/Drug Use subscale of the MAYSI-2 in self-rating by participants. The MAYSI-2 is a brief screening tool designed for youth between the ages of 12-17 years, but it has been suggested that the screening tool may also be adequate for young adults as long as results are interpreted with caution.
  The MAISY-2 contains 52 items across seven subscales: Alcohol/Drug Use, Anger-Irritability, Depression-Anxiety, Somatic Complaints, Suicide Ideation, Traumatic Experiences and Thought Disturbance. Respondents are asked about the presence of various thoughts, feelings or behaviours in the past few months, in a yes or no format. Each subscale contains different caution cut-offs.

OTHER OUTCOMES:
Client Training Satisfaction (2 intervention conditions) | T2 (post intervention, ≤2 weeks after end of intervention)
  Participants within the two intervention conditions can indicate their satisfaction with the training using the Client Satisfaction Questionnaire (CSQ) at T2 (post intervention). The CSQ was specifically developed to assess participants' experiences and satisfaction with START NOW. It contains eight items on a 4-point Likert-Scale (ranging from 0 to 3; response options are provided with smileys) and two open questions about what participants liked or would want to be changed within the training. Total scores can range from 0 to 24.
Trainer Satisfaction (facilitators of the group training) | T2 (post intervention, ≤2 weeks after end of intervention)
  Satisfaction of facilitators of the group training guided by a facilitator condition will be assessed with the Trainer Satisfaction Questionnaire (TSQ) at T2 (post intervention), a 5 Min self-rating questionnaire. After the end of the intervention, focused group discussions are planned for all interested institutions regarding implementation and experiences with START NOW. The group discussions will be conducted as guided interviews for 1 hour with a maximum of 3 institute employees and recorded for later transcription (audio and video; destroyed after transcription; text anonymized) and qualitative analyses.
Social Atmosphere | T1 and all following time points
  Social Atmosphere will be assessed by the German version of the Essen Climate Evaluation Schema (EssenCES). It is a short self-rating questionnaire, containing 17 items across three subscales: Therapeutic Hold, Patients' Cohesion and Mutual Support, and Experienced Safety. Responses are given on a 5-point Likert Scale (0= not at all, 1= little, 2= somewhat, 3= quite a lot, 4= very much). Total scores can range from 0 to 68 with higher scores indicating a better social climate. Accordingly, change scores can range between -68 to +68.
Checklist Baseline T1 and Checklist Monitoring | T1 and all following time points. NOTE: Monitoring purpose (Data Control), no aggregation of data
  Inclusion/exclusion criteria throughout the course of the study (i.e., participation in concurrent CBT based skills training similar to START NOW., internet access, external placements/discharge, unauthorized leaves) will be screened/monitored with two specially designed Checklists.
Prior Experiences of Caretakers and Facilitator | For caretakers at baseline (T1), for facilitators at post-treatment assessment (T2, ≤2 weeks after end of intervention).
  The professional qualification of involved caretakers and facilitators, their experiences with START NOW or other forms of resilience trainings will be assessed with a short questionnaire.
Adherence | during one session (either live or via online connection)
  For each institution, the quality of the group training guided by a facilitator will be rated by a START NOW facilitator during one session (either live or via online connection) using a Quality Assurance Form.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Stadler, Prof. Dr., Principal Investigator — University Psychiatric Clinics Basel
Locations (1):
- University Psychiatric Clinic, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kersten L, Pratzlich M, Mannstadt S, Ackermann K, Kohls G, Oldenhof H, Saure D, Krieger K, Herpertz-Dahlmann B, Popma A, Freitag CM, Trestman RL, Stadler C. START NOW - a comprehensive skills training programme for female adolescents with oppositional defiant and conduct disorders: study protocol for a cluster-randomised controlled trial. Trials. 2016 Dec 1;17(1):568. doi: 10.1186/s13063-016-1705-6. PMID 27903282
- [Background] Kersten L, Cislo AM, Lynch M, Shea K, Trestman RL. Evaluating START NOW: A Skills-Based Psychotherapy for Inmates of Correctional Systems. Psychiatr Serv. 2016 Jan;67(1):37-42. doi: 10.1176/appi.ps.201400471. Epub 2015 Aug 17. PMID 26278230
- [Background] Stadler C, Freitag CM, Popma A, Nauta-Jansen L, Konrad K, Unternaehrer E, Ackermann K, Bernhard A, Martinelli A, Oldenhof H, Gundlach M, Kohls G, Pratzlich M, Kieser M, Limprecht R, Raschle NM, Vriends N, Trestman RL, Kirchner M, Kersten L. START NOW: a cognitive behavioral skills training for adolescent girls with conduct or oppositional defiant disorder - a randomized clinical trial. J Child Psychol Psychiatry. 2024 Mar;65(3):316-327. doi: 10.1111/jcpp.13896. Epub 2023 Oct 10. PMID 37814906
- [Derived] Kersten L, Alfano J, Erlanger TE, Helfenstein F, Lanz L, Weiss S, Chilla C, von Planta B, Kapoor M, Borel N, Rocco T, Papageorgiou A, De Brito CF, Bajrami A, Savary V, Mayor M, Hurschler J, Traut A, Brunner D, Vriends N, Stadler C. START NOW WebApp-promoting emotion regulation and resilience in residential youth care and correctional institutions: study protocol for a cluster randomized controlled trial. Trials. 2024 May 22;25(1):341. doi: 10.1186/s13063-024-08180-z. PMID 38778383